CLINICAL TRIAL: NCT01444911
Title: Evaluation of a Multifaceted Vaginal Renewal™ Program Utilizing Vibrating Wands in Gynecologic Cancer Patients Experiencing Sexual Dysfunction: A Randomized Controlled Trial
Brief Title: Evaluation of The Vaginal Renewal™ Program in Gynecologic Cancer Patients Experiencing Sexual Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0217; OS10706 (Other: University of Wisconsin Carbone Cancer Center); NCI-2011-03674 (Registry Identifier: NCI Trial ID); A532820 (Other: UW Madison); SMPH\OBSTET & GYNEC\GYNEC ONC (Other: UW Madison)
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-07

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Sexual Dysfunction; Gynecologic cancer; Cancer survivor; Vaginal dilator
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Renewal Program (Experimental)
  Interventions: Device: Vaginal Renewal Program
- Standard of care (Active Comparator): This will consist of still vaginal dilator and/or lubricant.
  Interventions: Device: Vaginal Dilator

INTERVENTIONS:
Device: Vaginal Renewal Program — The Vaginal Renewal™ Program (VRP) consists of instructions on the use of a vibrating vaginal wand along with a particular water based lubricant.
  Arms: Vaginal Renewal Program
Device: Vaginal Dilator — Still vaginal dilator with lubricant.
  Arms: Standard of care

SUMMARY:
This is a randomized controlled trial designed to evaluate the effect of the Vaginal Renewal™ Program (VRP), consisting of the use of a vibrating vaginal wand, manual massage and a water based lubricant, on sexual dysfunction, compared to the current standard care for women with no evidence of disease after treatment for gynecologic cancers.

In the University of Wisconsin gynecologic oncology and radiation oncology clinics, patients are generally asked about sexual function. Those women who report sexual dysfunction will be given the option to enroll in the study. After enrollment, the Female Sexual Function Index (FSFI) and other quality of life surveys will be administered at baseline. The participants will be randomized to either the control arm, composed of standard of care therapy for the physical components of sexual dysfunction, or the experimental arm (VRP).

Throughout the study, the participants will undergo physical exams to assess the rate of improvement in their comfort with pelvic exams and changes in vaginal length. They will also be evaluated with the FSFI, Marinoff Scale for Dyspareunia, and Functional Assessment of Cancer Therapy-General (FACT-G) surveys at the end of the study to assess the magnitude of improvement in sexual function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* History of a gynecologic cancer
* No evidence of disease at time of inclusion in the study
* Postmenopausal (either surgical or natural menopause)
* Self report of sexual dysfunction that did not predate cancer diagnosis
* Suspected physical component to sexual dysfunction with the participant, not sexual partner
* Desire to improve sexual function
* ECOG Performance status score of 2 or better
* Six months or greater from last surgical and/or radiation treatment

Exclusion Criteria:

* History of sexual reassignment
* Presence of vaginal fistula
* Does not desire to improve sexual function
* Already using the vaginal renewal program
* Not fluent in English
* Incarceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health Madison, Wisconsin, United States, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a history of a gynecologic cancer and self-reported sexual dysfunction that was new or worsened since cancer diagnosis, and were randomized to one of two arms. All participants enrolled at the Gynecologic Oncology and Radiation Oncology clinics at the University of Wisconsin Carbone Cancer Center.
Period: Overall Study
Arm/Group | Vaginal Renewal Program | Standard of Care
Started | 16 | 13
Completed | 8 | 13
Not Completed | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Renewal Program | Standard of Care | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29
Pelvic Radiation [Number; unit: participants]
  Prior Pelvic Radiation | 2 | 1 | 3
  No Prior Pelvic Radiation | 14 | 12 | 26
Primary Disease Site [Number; unit: participants]
  Ovary | 5 | 5 | 10
  Endometrium | 6 | 6 | 12
  Cervix | 3 | 1 | 4
  Vulva | 1 | 0 | 1
  Dual Primary (Ovary and Endometrium) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Female Sexual Function Index (FSFI) Score at 6 Months
Description: Female Sexual Function Index (FSFI), uses a 19-item sexual functioning questionnaire to rate sexual function between 2.0 and 36.0, where 2.0 is low sexual function and 36.0 is high sexual function. Difference in FSFI scores are reported.
Time Frame: At baseline and 6 months
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Vaginal Renewal Program | Standard of Care
Number analyzed (Participants) | 8 | 13
Units on a scale | 5.575 [-8.4 to 14] | 6.069 [-4.0 to 20.8]
Statistical Analysis 1: Comparison: Vaginal Renewal Program vs Standard of Care; Test type: Superiority or Other; p = 0.89, ANOVA

2. Secondary Outcome: Change in Marinoff Scale at 6 Months
Description: The Marinoff dyspareunia scale measures pain with intercourse, measured from 0-3, according to the following scale:
  0 = no pain with intercourse
  1. = pain with intercourse that doesn't prevent the completion
  2. = pain with intercourse requiring interruption or discontinuance
  3. = pain with intercourse preventing any intercourse
  Difference in Marinoff scores reported, value at 6 months minus value at baseline.
Time Frame: At baseline and 6 months
Population: Data for eleven subjects (2 from Standard of Care and 9 from VRP) was not collected at one or more study visits, and the change in scores could not be calculated.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vaginal Renewal Program | Standard of Care
Number analyzed (Participants) | 7 | 11
units on a scale | -0.857 [-2 to 0] | -0.818 [-3 to 0]

3. Secondary Outcome: FACT-G Score
Description: The FACT-G (Functional Assessment of Cancer Therapy - General) questionnaire assesses general cancer quality-of-life measure for evaluating patients receiving cancer treatment. Scores range from 0 to 108, where 0 is low well-being and 108 is the highest well-being possible. Difference in score from baseline to 6 months is reported.
Time Frame: At baseline and 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vaginal Renewal Program | Standard of Care
Number analyzed (Participants) | 8 | 13
units on a scale | 4.375 [-15 to 22] | 4.872 [-1 to 25]

4. Secondary Outcome: Vaginal Length
Description: Change in vaginal length as measured from baseline to 6 months.
Time Frame: At baseline and 6 months
Measure: Mean (Full Range); unit: Centimeters
Arm/Group | Vaginal Renewal Program | Standard of Care
Number analyzed (Participants) | 8 | 13
Centimeters | 1.188 [0 to 3.5] | 0.154 [-3 to 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year, 8 months.
Description: Participants were assessed for toxicity at each study visit. All events at least possibly related to the study intervention will be collected. Participants were instructed to call the study team for adverse events that occurred between visits. The study team or an on-call physician were available 24 hours a day.
Arm/Group | Vaginal Renewal Program | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 4/16 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Renewal Program (N=16) | Standard of Care (N=13)
Bladder irritation (Renal and urinary disorders) | 1 (1) | 0
Bladder pressure (Renal and urinary disorders) | 1 (1) | 0
Urinary tract infections (UTI) (Infections and infestations) | 1 (1) | 2 (3)
Vaginal infection (Reproductive system and breast disorders) | 1 (1) | 0 — Yeast
Vaginal irritation (Reproductive system and breast disorders) | 1 (1) | 0
Vulvar fissures (Reproductive system and breast disorders) | 1 (1) | 0
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed before completion due to a slowing accrual rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No